CLINICAL TRIAL: NCT06677580
Title: Multidisciplinary Network OSA Code (Obstructive Apnea Syndrome): Digital Operative Model in Public Health for an Early Diagnosis and Therapy Monitoring, a Monocentric Observational Prospective Study
Brief Title: Multidisciplinary Network OSA Code (Obstructive Apnea Syndrome): Digital Operative Model in Public Health for an Early Diagnosis and Therapy Monitoring
Acronym: DOMOSA
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Luigi Ferini Strambi, Prof, IRCCS San Raffaele
Other Study IDs: CET 94-2023
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: OSA - Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) is a sleep related breathing disorder with high epidemiological impact (9-38% of general population), more frequently reported in male gender and increasing with the age. Pathognomonic OSAS symptoms are snoring, excessive daytime sleepiness, sleep fragmentation, awakening during the night often for nocturia and morning headache. The repeated sleep fragmentation due to numerous awakenings (the patient is often unaware of this) can impair higher cognitive functions over the time and negatively impact the quality of life, If timely untreated.

Among the most frequently impaired cognitive functions detected in OSAS patients, there are attention, concentration, amnestic and executive domains. While these impairments are well documented in literature, the pathogenetic mechanisms underlying cognitive impairment are not yet defined. To date, the most widely accepted pathophysiological hypotheses are two: i) intermittent hypoxia (frequent brain awakenings); ii) sleep fragmentation. Moreover solid evidence report that, there is a strict correlation between OSAS and neurodegenerative diseases, such as Mild Cognitive Impairment (MCI) and Alzheimer's Dementia (AD). Indeed, OSAS might act as a trigger, accelerating the accumulation of harmful proteins in the brain, in particular beta-amyloid and tau protein.

The first-line treatment for OSAS is Continuous Positive Airway Pressure (CPAP). Of note is the effect of CPAP treatment on higher cognitive function in OSAS patients.

Not all OSAS' patients, however, develop MCI/AD over time. For this reason, to identify the OSA phenotype (both clinical and neuroimaging) at higher risk of phenoconversion represents an important challenge for neuropsychologists and neurologists.

The interest on OSAS is not purely scientific, but also economic, whit important repercussions on the intake and costs of hospital and home management of OSAS' patients.

In conclusion, OSAS is a syndrome needing great attention for several reasons: i) from a scientific point of view, it is important to identify for the risk of phenoconversion to highly disabling neurodegenerative diseases; ii) from an economic-welfare point of view, to reduce costs that still burden NHS.

In summary, the study may have an important impact on Public Health, considering the various aspects related to the taking care and management of OSAS' patients: 1) To know in details, the syndrome epidemiology and on this basis provide for the corresponding commitment of resources, suitable for implementing the support activities for both patients and families; 2) To have major information on the real prevalence of clinical signs and symptoms, to support and optimize the care efforts of physicians; 3) To assess the prognostic factors and outcomes of the treatment; 4) On the basis of the data collected in the platform, to have the possibility for support research.

OSAS-platform could represent one of the most effective methods to improve scientific, clinical and therapeutical knowledge on OSAS-pathology.

ELIGIBILITY:
Inclusion Criteria:

* patients with obstructive sleep apnea syndrome (Diagnosis according to American Academy of Sleep Society International Classification of Sleep Disorders, third edition (ICSD-3))
* male and female
* age > 18 years

Exclusion Criteria:

* Unable of giving signed informed consent
* Refuse to participate or withdrawal the consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patientswith obstructive sleep apnea syndrome, male and female, with age > 18 years
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
To characterize the profile of patients with obstructive sleep apnea syndrome (afferent to IRCCS San Raffaele Hospital, UO Neurology - Sleep Disorders Center, Milan) at higher risk of conversion to neurodegenerative diseases | From enrollment to the end of 3 years of follow-up
  To characterize the profile of patients with obstructive sleep apnea syndrome (afferent to IRCCS San Raffaele Hospital, UO Neurology - Sleep Disorders Center, Milan) at higher risk of conversion to neurodegenerative diseases, particularly Alzheimer's Dementia and Mild Cognitive Impairment

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele Hospital - Sleep Disorders Center, Milan, Italy, Italy